CLINICAL TRIAL: NCT02723929
Title: Effects of Transcranial Direct Current Stimulation (tDCS) and Transcranial Ultrasound (TUS) on the Perception of Pain and Functional Limitations Due to Osteoarthritis of the Knee
Brief Title: Effects of tDCS and tUS on Pain Perception in OA of the Knee
Status: Active, not recruiting | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P000486
Record Dates: First submitted 2016-02-26; First posted 2016-03-31 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Osteoarthritis
Keywords: transcranial direct current stimulation; transcranial ultrasound; non-invasive brain stimulation
MeSH Terms: conditions — Chronic Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: tDCS and tUS
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Active Electrical Stim/Active Ultrasound (Experimental): Subjects will undergo active low-intensity transcranial electrical stimulation in conjunction with active transcranial ultrasound for 20 minutes.
  Interventions: Device: active low-intensity transcranial electrical stimulation/active transcranial ultrasound
- Sham Electrical Stim/Sham Ultrasound (Sham Comparator): Subjects will undergo sham (placebo) low-intensity transcranial electrical stimulation in conjunction with sham transcranial ultrasound for 20 minutes.
  Interventions: Device: Sham low-intensity transcranial electrical stimulation/sham transcranial ultrasound

INTERVENTIONS:
Device: active low-intensity transcranial electrical stimulation/active transcranial ultrasound — Subjects will undergo 20 minutes of low-intensity transcranial electrical stimulation of up to 2mA. During active stimulation, the current will be active for the full 20 minutes.
  Subjects will also undergo 20 minutes of transcranial ultrasound. During active stimulation, the ultrasound will be active for the full 20 minutes.
  Arms: Active Electrical Stim/Active Ultrasound
Device: Sham low-intensity transcranial electrical stimulation/sham transcranial ultrasound — Subjects will undergo 20 minutes of low-intensity transcranial electrical stimulation, as in the active condition; however, during sham stimulation (placebo) the current will not be active for the full 20 minutes.
  Subjects will also undergo 20 minutes of transcranial ultrasound in the same par. During active stimulation, the ultrasound will be active for 20 minutes - however, during sham stimulation (placebo) the ultrasound will not be active for the full 20 minutes.
  Arms: Sham Electrical Stim/Sham Ultrasound

SUMMARY:
The purpose of this study is to investigate the effects of transcranial direct current stimulation (tDCS) in conjunction with transcranial ultrasound (TUS) on pain perception and functional limitations in people with osteoarthritis of the knee. The investigators hypothesize that there will be a decrease in pain levels with active stimulation, when compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study.
2. Subjects between 18-85 years old.
3. Diagnosis of chronic osteoarthritis with pain of either knee as self-reported.
4. Existing knee pain of at least 3 on a 0-10 VAS scale on average over the past 6 months.
5. Pain of at least 3 on a 0-10 VAS scale on average over the week prior to the first stimulation session.
6. Pain resistant to common analgesics and medications for chronic pain used as initial pain management such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex, and Codeine.
7. Having the ability to feel pain as self-reported.

Exclusion Criteria:

1. Pregnancy or trying to become pregnant in the next 6 months.
2. History of alcohol or drug abuse within the past 6 months as self-reported
3. Contraindications to transcranial brain stimulation or TUS, i.e. implanted brain medical devices or implanted brain metallic devices.
4. Unstable medical conditions (e.g. uncontrolled diabetes, uncompensated cardiac issues, heart failure or chronic obstructive pulmonary disease).
5. Epilepsy.
6. Use of carbamazepine within the past 6 months as self-reported.
7. Suffering from severe depression (with a score of >30 in the Beck Depression Inventory)
8. History of unexplained fainting spells as self-reported.
9. Head injury resulting in more than a momentary loss of consciousness
10. History of neurosurgery as self-reported.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2026-12-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Network Research Institute, Charlestown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 64 subjects were enrolled and randomized
Groups:
- Active Electrical Stim/Active Ultrasound: Subjects will undergo active low-intensity transcranial electrical stimulation in conjunction with active transcranial ultrasound for 20 minutes.
  Active low-intensity transcranial electrical stimulation/active transcranial ultrasound: Subjects will undergo 20 minutes of low-intensity transcranial electrical stimulation. During active stimulation, the current will be active for the full 20 minutes.
  Subjects will also undergo 20 minutes of transcranial ultrasound. During active stimulation, the ultrasound will be active for the full 20 minutes.
- Sham Electrical Stim/Sham Ultrasound: Subjects will undergo sham (placebo) low-intensity transcranial electrical stimulation in conjunction with sham transcranial ultrasound for 20 minutes.
  Sham low-intensity transcranial electrical stimulation/sham transcranial ultrasound: Subjects will undergo 20 minutes of low-intensity transcranial electrical stimulation, as in the active condition; however, during sham stimulation (placebo) the current will not be active for the full 20 minutes. Subjects will also undergo 20 minutes of transcranial ultrasound. During active stimulation, the ultrasound will be active for 20 minutes - however, during sham stimulation (placebo) the ultrasound will not be active for the full 20 minutes.
Period: Overall Study
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Started | 30 | 34
Completed | 24 | 24
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Population: Baseline participants for randomized subjects
Groups:
- Active Electrical Stim/Active Ultrasound: Subjects will undergo active low-intensity transcranial electrical stimulation in conjunction with active transcranial ultrasound for 20 minutes.
  active low-intensity transcranial electrical stimulation/active transcranial ultrasound: Subjects will undergo 20 minutes of low-intensity transcranial electrical stimulation of up to 2mA. During active stimulation, the current will be active for the full 20 minutes.
  Subjects will also undergo 20 minutes of transcranial ultrasound. During active stimulation, the ultrasound will be active for the full 20 minutes.
- Sham Electrical Stim/Sham Ultrasound: Subjects will undergo sham (placebo) low-intensity transcranial electrical stimulation in conjunction with sham transcranial ultrasound for 20 minutes.
  Sham low-intensity transcranial electrical stimulation/sham transcranial ultrasound: Subjects will undergo 20 minutes of low-intensity transcranial electrical stimulation, as in the active condition; however, during sham stimulation (placebo) the current will not be active for the full 20 minutes.
  Subjects will also undergo 20 minutes of transcranial ultrasound in the same par. During active stimulation, the ultrasound will be active for 20 minutes - however, during sham stimulation (placebo) the ultrasound will not be active for the full 20 minutes.
- Total: Total of all reporting groups
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound | Total
Number analyzed (Participants) | 30 | 34 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.4) | 61.8 (8.7) | 61.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 34 | 64

OUTCOME MEASURES:

1. Primary Outcome: Changes in Pain Scale as Measured by VAS
Description: Changes in the Visual Analogue Scale (VAS) for pain were measured in order to determine whether transcranial direct current stimulation in conjunction with transcranial ultrasound is effective in reducing pain in subjects with Osteoarthritis of the Knee.
  The VAS scale goes from 0 up to 10, where 0 means no pain at all and 10 means the worst imaginable pain and is reported following the full course of therapy. Since we are using a difference, smaller values (negative) represent a better outcome
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Number analyzed (Participants) | 30 | 34
units on a scale | -2.21 (0.2) | -1.6 (0.1)

2. Secondary Outcome: Average Daily Dose of Acetaminophen Equivalent
Description: Analgesic use (average daily dose of acetaminophen equivalent)
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Acetaminophen equivalent in mg
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Number analyzed (Participants) | 30 | 34
Acetaminophen equivalent in mg | 390.7 (47.1) | 1116.4 (98.6)

3. Secondary Outcome: Changes in Pain Scale as Measured by VAS
Description: Changes in the Visual Analogue Scale (VAS) for pain were measured in order to determine whether transcranial direct current stimulation in conjunction with transcranial ultrasound is effective in reducing pain in subjects with Osteoarthritis of the Knee.
  The VAS scale goes from 0 up to 10, where 0 means no pain at all and 10 means the worst imaginable pain. Since we are using a difference, smaller values (negative) represent a better outcome.
Time Frame: Baseline and 4 weeks post-stimulation
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Number analyzed (Participants) | 30 | 34
units on a scale | -2.91 (0.38) | -1.28 (0.30)

4. Secondary Outcome: Percentage Change in Diffuse Noxious Inhibitory Controls (DNIC) From Baseline
Description: This measures the endogenous pain modulatory pathway. This study will evaluate DNIC in pain patients using pressure as the test stimulus, and cold water as the conditioning stimulus. DNIC will be induced approximately 1-min later by having subjects immerse their hand into a water bath maintained at 10-12˚C for approximately 1 min. Parallel to the last 30s of DNIC conditioning (cold water immersion), the pressure test stimulus will be reapplied. DNIC response will be calculated as the difference between the average of pain ratings from the test stimulus minus the average of pain ratings during the conditioned stimulus. Larger percentage change means a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Number analyzed (Participants) | 30 | 34
Percentage change from baseline | 12 (2.9) | 4.0 (1.8)

5. Secondary Outcome: Percentage Change From Baseline in the Single Leg Standing Balance Test
Description: We will record the time (seconds) for which a subject is able to stand unsupported on one foot while looking straight ahead with hands on hips. Larger percentage change means a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Number analyzed (Participants) | 30 | 34
Percentage change from baseline | 17.5 (4.5) | 3.0 (3.1)

6. Secondary Outcome: Percentage Change From Baseline in the Step Test
Description: The subject was asked to stand unsupported with their feet parallel to each other in front of a step. We assessed the number of times the participant could place their foot up onto the step and return it to the floor over a 15-sec interval. Larger percentage change means a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Number analyzed (Participants) | 30 | 34
Percentage change from baseline | 27.0 (2.0) | 18.7 (1.8)

7. Secondary Outcome: Percentage Change in Functional Reach Test From Baseline
Description: Subject will be instructed to stand next to, but not touch the wall, and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist. Smoothness of wrist movement is assessed as the subject was asked to outstretch their arm in a maximal forward reach, while maintaining a fixed base of support. Smoothness is dimensionless and is calculated as mean speed divided by peak speed. Larger percentage change means a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
Number analyzed (Participants) | 30 | 34
Percentage change from baseline | 12.4 (2.8) | 3.3 (2.3)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Adverse effects were collected with a questionnaire for adverse effects
Arm/Group | Active Electrical Stim/Active Ultrasound | Sham Electrical Stim/Sham Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/34
Other Adverse Events (participants affected / at risk) | 23/30 | 29/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Electrical Stim/Active Ultrasound (N=30) | Sham Electrical Stim/Sham Ultrasound (N=34)
Tingling (Nervous system disorders) | 23 | 29 — Sensation of tingling near the stimulation site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT02723929/Prot_SAP_000.pdf